CLINICAL TRIAL: NCT03379623
Title: A Feasibility Randomised Controlled Trial of the Implementation in Malaysian Healthcare Context of the ESCAPE-pain Programme for Patients With Knee Osteoarthritis
Brief Title: ESCAPE-pain Programme in Malaysia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Kamil Che Hasan (Other)
Responsible Party: Sponsor-Investigator, Muhammad Kamil Che Hasan, PhD Candidate, University of Manchester
Organization: University of Manchester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017-2045-3627
Record Dates: First submitted 2017-11-28; First posted 2017-12-20 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomization will be performed by an independent person from Kulliyyah of Nursing research unit. The researcher will not be involved in allocation to intervention or control group. The participants will be advised not to talk about the study during assessments to prevent unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: ESCAPE-pain Programme
- Usual care group (No Intervention)

INTERVENTIONS:
Other: ESCAPE-pain Programme — The Enabling Self-management and Coping with Arthritic (knee) Pain using Exercise (ESCAPE-pain) is a programme of rehabilitation that integrates educational self-management and coping strategies for people with joint pain with an individualised exercise regimen for each participant. The implementation of the programme will be conducted by the researcher as a certified facilitator by using Clinician's training manual for the ESCAPE-pain programme.
  Arms: Intervention group

SUMMARY:
The overall aim of this study is to develop an evidence based exercise programme for the management of knee osteoarthritis which is feasible and acceptable to patients and healthcare professionals in Malaysia. The chosen programme was identified through a systematic literature search and is the programme developed by Hurley et al. in 2007. This programme will be evaluated through mixed-methods sequential exploratory design research study guided by the United Kingdom (UK) Medical Research Council guidance and framework. It involves two phases of data collection. The first phase (already completed) comprised a qualitative study aimed at exploring the beliefs and attitudes of Malaysian people that would need to be taken into account when adapting the evidence based ESCAPE-pain (acronym for 'Enabling Self-management and Coping with Arthritic pain using Exercise) programme for implementation in the context of Malaysian healthcare system. The second phase will be conducted to evaluate the feasibility of trialling ESCAPE-pain programme in Malaysia.

DETAILED DESCRIPTION:
In Malaysia, functional limitations and impaired daily living activities affect patients with knee osteoarthritis (OA) in such a way that they tend to refrain from hospital visits. This may may lead to depression and reduced quality of life, which may then impact on increases in health care costs. The service provided by hospitals to these patients, is under-utilised by the multi-ethnic people that make up the population. Through the researcher's previous clinical experience, it was observed that patients were complaining of difficulty in getting to the hospital, long waiting times, and also increasing transport costs. Thus, adoption of self-care and early prevention has been suggested as a solution for the OA affected Malaysian community. In addition, there is no home based exercise programme for patients with knee OA in current health practice in Malaysia. Although some of these patients in Malaysia are prescribed with home-based exercises, a fully comprehensive self-management programme is lacking for patients generally. Therefore, there is a need for a home based self-management exercise programme for people with knee OA which can be implemented in community setting without frequent involvement of the hospitals. The UK Medical Research Council Guidance and Framework on developing and evaluating complex interventions will be used to facilitate the process of developing a complex intervention. A systematic review of the literature identified an exercise programme called ESCAPE-Pain as the programme with the best evidence for adaptation as a self-management programme to implement in Malaysia.

In phase 1, (already conducted), the investigators have undertaken interviews with patients and healthcare professionals (HCPs) in Malaysia to identify their beliefs and attitudes towards the ESCAPE-pain programme. Preliminary analysis reveals that patients with knee OA and HCPs have positive views towards the implementation of the programme with integration of a few new components.

In this phase, the investigators propose to undertake a feasibility randomised controlled trial in which the investigators compare the modified ESCAPE-pain programme for the Malaysian context, versus usual care in Malaysian OA patients. ESCAPE-pain is a rehabilitation programme that helps people with osteoarthritis (OA) and/or chronic joint pain to self -manage their condition. The programme aims to increase physical function and improve quality of life. The ESCAPE-pain programme, will be run over six weeks, with participants attending for one hour session, twice a week. Each session contains around a 20 minutes themed discussion focused on helping to support self-management and followed by about 45 minutes of exercise. The sessions will be led by the researcher who trained in how to deliver the ESCAPE-pain programme.

This feasibility study is required to identify the best methods for a definitive trial in the future, to test recruitment and other trial procedures, the acceptability of the intervention and the way it is implemented and to provide insight into appropriateness of our outcome measures, including providing data to permit estimation of effect size to be used in sample size calculations for a definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older (one of the criteria to diagnose knee osteoarthritis by a medical officer based on Ministry of Health Malaysia guidelines (MoH, 2014)).
* Diagnosed with osteoarthritis affecting the knee by medical officer based on Clinical Practice Guidelines (CPG) MOH (MOH, 2014).
* Independently mobile either with or without walking aid.
* Approved medically fit for exercise by a medical officer.
* Able to communicate in Malay language.
* Must have mental capacity to give informed consent.

Exclusion Criteria:

* Had knee replacement / lower limb arthroplasty.
* Intraarticular injections within past six months.
* Have any significant musculoskeletal issues (e.g. inflammatory arthritis, connective tissue diseases, fibromyalgia, severe osteoporosis, peripheral neuropathy, or gout).
* Very severe joint pain which limiting mobility to less than 50 metres.
* people with unstable co-morbidities (such as cardiovascular and respiratory conditions, type 2 diabetes, severe pain in other joints).
* wheelchair user.
* severe cognitive impairment assessed by a medical officer.
* severe auditory or visual impairment assessed by a medical officer.
* inability to comprehend the ESCAPE-pain procedure

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline The Knee Injury and Osteoarthritis Outcome Score (KOOS) at 6 and 12 weeks | Baseline, after intervention completion at week 6, and at week 12 of intervention for follow-up.
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient-reported outcome measurement instrument, developed to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.

SECONDARY OUTCOMES:
Change of Baseline Timed up and Go Test at 6 and 12 weeks | Baseline, after intervention completion at week 6, and at week 12 of intervention for follow-up.
  The purpose is to measure lower limb strength and balance while moving. A chair will be placed next to a wall and the marker 8 feet will be marked with a cone in front of the chair. The path between the chair and the marker will be cleared from any obstacle. The participant will be started with fully seated with hands resting on the knees and feet flat on the ground. On the command, "Go," timing will be started and the subject stands and walks (no running) as quickly as possible (and safely) to and around the cone, returning to the chair to sit down. The time will be stopped as they sit down. It will be performed two trials. Participants will be given a chance to do practice trial before actual time measured. The average time will be recorded to the nearest 1/10th second.
Change of Baseline Health Beliefs and Self-efficacy for exercise at 6 and 12 weeks | Baseline, after intervention completion at week 6, and at week 12 of intervention for follow-up.
  A simple outcome measure that captures the benefit people attain from exercise. It is by altering their ability to exercise effectively and their beliefs towards exercise.A 17-items questionnaires to reflect the beliefs about one's ability to exercise (self-efficacy for exercise) (4 items), barriers to exercise (3 items), benefits of exercise (3 items), and impact of exercise on arthritis (7 items). The items use a 5-point Likert scale, ranging from strongly agree to strongly disagree, to indicate their beliefs.
Change of Baseline The Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) at 6 and 12 weeks | Baseline, after intervention completion at week 6, and at week 12 of intervention for follow-up.
  SWEMWBS is used in the context of projects and programmes to enable self-reflection as a prelude to involvement with health enhancing activities. It does seem to be sensitive to changes in mental wellbeing at the individual level. Each of the 7 statement responses in SWEMWBS are scored from 1 to 5, from 'none of the time' to 'all of the time'. A total score is calculated by summing the 7 individual statement scores. The minimum score is 7 and the maximum is 35.
Change of Baseline Short Falls Efficacy Scale-International (FES-I) at 6 and 12 weeks | Baseline, after intervention completion at week 6, and at week 12 of intervention for follow-up.
  The short Falls Efficacy Scale-International (FES-I) is a validated and reliable 7-item tool which measures confidence in performing a range of activities of daily living without falling. This scale has recently been modified to maximise its suitability for a range of different languages and cultures (Yardley et al. 2005). Participants will be asked to rate, on a four-point Likert scale,their concerns about the possibility of falling when performing 7 activities. Participants will be instructed to rate each activity regardless of whether they actually perform it. The scores are added up to calculate a total score that ranges from 7 to 28 for the short FES-I. A higher score indicates a greater fear of falling.
Exercise Adherence Rating Scale (EARS) | Week 12 of intervention
  Exercise Adherence Rating Scale (EARS) is an assessment measuring tool to assess adherence to prescribed home exercise. It consists of 6 statements that best describes how participants do their recommended exercises/activities. The EARS is scored on a 5-point Likert scale (0 - completely agree to 4 - completely disagree). Items 1, 4 and 6 are reverse scored, resulting in a possible score of between 0 and 24. A higher score indicates better adherence.

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - IIUM Medical Centre, Kuantan, Pahang

REFERENCES:
- [Background] Hurley MV, Walsh NE, Mitchell HL, Pimm TJ, Patel A, Williamson E, Jones RH, Dieppe PA, Reeves BC. Clinical effectiveness of a rehabilitation program integrating exercise, self-management, and active coping strategies for chronic knee pain: a cluster randomized trial. Arthritis Rheum. 2007 Oct 15;57(7):1211-9. doi: 10.1002/art.22995. PMID 17907147
- [Background] Hurley MV, Walsh NE, Mitchell HL, Pimm TJ, Williamson E, Jones RH, Reeves BC, Dieppe PA, Patel A. Economic evaluation of a rehabilitation program integrating exercise, self-management, and active coping strategies for chronic knee pain. Arthritis Rheum. 2007 Oct 15;57(7):1220-9. doi: 10.1002/art.23011. PMID 17907207
- [Background] Jessep SA, Walsh NE, Ratcliffe J, Hurley MV. Long-term clinical benefits and costs of an integrated rehabilitation programme compared with outpatient physiotherapy for chronic knee pain. Physiotherapy. 2009 Jun;95(2):94-102. doi: 10.1016/j.physio.2009.01.005. Epub 2009 Mar 21. PMID 19627690
- [Background] Hauer KA, Kempen GI, Schwenk M, Yardley L, Beyer N, Todd C, Oster P, Zijlstra GA. Validity and sensitivity to change of the falls efficacy scales international to assess fear of falling in older adults with and without cognitive impairment. Gerontology. 2011;57(5):462-72. doi: 10.1159/000320054. Epub 2010 Oct 22. PMID 20975251
- [Background] Newman-Beinart NA, Norton S, Dowling D, Gavriloff D, Vari C, Weinman JA, Godfrey EL. The development and initial psychometric evaluation of a measure assessing adherence to prescribed exercise: the Exercise Adherence Rating Scale (EARS). Physiotherapy. 2017 Jun;103(2):180-185. doi: 10.1016/j.physio.2016.11.001. Epub 2016 Nov 9. PMID 27913064
- [Background] Zulkifli MM, Kadir AA, Elias A, Bea KC, Sadagatullah AN. Psychometric Properties of the Malay Language Version of Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire among Knee Osteoarthritis Patients: A Confirmatory Factor Analysis. Malays Orthop J. 2017 Jul;11(2):7-14. doi: 10.5704/MOJ.1707.003. PMID 29021872
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398